CLINICAL TRIAL: NCT06411522
Title: Clinical and Microbiological Comparison Between 0.12% Chlorhexidine and 0.05% Chlorhexidine + 0.05% Cetylpyridinium Chloride Mouthwashes in Chemical Biofilm Control During Supportive Periodontal Therapy: A Randomized Clinical Study
Brief Title: Clinical and Microbiological Comparison of 0.12% CHX and 0.05% CHX+0.05%CPC Mouthwashes in TPS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Nicola Discepoli, Professor, University of Siena
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Perio_Micro_01
Record Dates: First submitted 2024-05-01; First posted 2024-05-13 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Chlorhexidine; Gingivitis; Periodontitis; Cetylpyridinium Chloride
Keywords: Prevention
MeSH Terms: conditions — Gingivitis; Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Test 1 (Active Comparator): Following the completion of a comprehensive periodontal charting, and prior to assigning the patient to one of the two experimental groups, patients will undergo an Oral Hygiene Instruction and Motivation (OHIM) session using a manual toothbrush, individualized interdental brushes, and a commercially available toothpaste containing sodium fluoride. Subsequently, a professional mechanical plaque removal (PMPR) will be performed by the operator, consisting of a conventional dental hygiene session.
  In treatment Test 1 patients will receive mouthwash containing 0.12% CHX (Chlorhexidine). Each patient will be instructed to use the assigned mouthwash twice a day (15 ml for 30 s) after common practices of home oral hygiene. Follow-up visits will occur at 1, 2, 3, and 6 months, during which participants will be clinically examined. Microbiological samples will be collected at 1, 2, and 3 months.
  Interventions: Device: Mouthwash containing 0.12% CHX (Chlorhexidine)
- Treatment Test 2 (Experimental): After completing a thorough periodontal charting and before allocating patients to one of the two experimental groups, they will receive an Oral Hygiene Instruction and Motivation (OHIM) session using a manual toothbrush, personalized interdental brushes, and a commercially available toothpaste containing sodium fluoride. Following this, an operator will conduct a professional mechanical plaque removal (PMPR), which entails a standard dental hygiene procedure.
  In Treatment Test 2 patients will receive mouthwash containing 0.05% CHX (Chlorhexidine) and 0.05% CPC (Cetylpyridinium Chloride) as the main active ingredients in a patented formulation with optimized bioavailability and they will be instructed to use it twice daily (15 ml for 30 s) following their regular home oral hygiene routine.
  Follow-up appointments will be scheduled at 1, 2, 3, and 6 months for clinical examinations of participants, with microbiological samples being collected at 1, 2, and 3 months.
  Interventions: Device: Mouthwash containing 0.05% CHX (Chlorhexidine) and 0.05% CPC (Cetylpyridinium Chloride)

INTERVENTIONS:
Device: Mouthwash containing 0.12% CHX (Chlorhexidine) — Following the execution of a full mouth periodontal chart, the delivery of oral hygiene instructions and motivation and a session of full mouth ultrasonic debridement, patients, according to the allocation group, will receive a 0.2% CHX mouthwash. Patients will be instructed to use the delivered mouthwashes twice a day (15 ml for 30 seconds).
  Arms: Treatment Test 1
Device: Mouthwash containing 0.05% CHX (Chlorhexidine) and 0.05% CPC (Cetylpyridinium Chloride) — Following the execution of a full mouth periodontal chart, the delivery of oral hygiene instructions and motivation and a session of full mouth ultrasonic debridement, patients, according to the allocation group, will receive a 0.05% CHX + 0.05% CPC mouthwash. Patients will be instructed to use the delivered mouthwashes twice a day (15 ml for 30 seconds).
  Arms: Treatment Test 2

SUMMARY:
The present study compares the effectiveness of two mouthwash formulations (0.12% CHX and 0.05% CHX+0.05%CPC) in reducing gingival inflammation and microbial colonization in individuals with gingivitis and in preventing periodontitis recurrence. The main focus is on assessing the clinical impact of the mouthwashes over six months, with a secondary goal of evaluating their effect on systemic blood pressure.

DETAILED DESCRIPTION:
This study aims to assess the impact of at-home use of 0.05% CPC + 0.05% chlorhexidine or 0.12% chlorhexidine, combined with professional plaque removal, on gingival inflammation and microbial quantity and quality in individuals diagnosed with gingivitis and reduced periodontium. It seeks to identify the most effective mouthwash formulation for reducing microbial colonization and preventing periodontitis recurrence. Comparing the commonly used 0.12% chlorhexidine with the alternative formulation of 0.05% chlorhexidine + 0.05% CPC over one month, with no reported side effects, is the main focus. The study does not pose risks to participants, with the main inconvenience being tooth enamel darkening, which can be easily resolved with professional dental cleaning. The primary objective is to evaluate the additional clinical effect of both formulations after professional plaque removal over six months in patients undergoing supportive periodontal therapy. The secondary objective is to assess the impact of these antimicrobials on systemic blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Bleeding on probing (BOP) ≥10%,
* No more than 4 sites with pocket depth (PPD) >5mm
* Presence of attachment loss (AL) and radiographic bone loss (RBL)
* A minimum of 20 teeth

Exclusion Criteria:

* Intolerance or allergy to antimicrobials
* Systemic therapy with anticoagulants/beta-blockers
* Local/systemic antibiotic therapy 3 months before
* Inability to understand and sign the written informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-10-18 (Actual); Study Completion 2025-10-18 (Actual)

PRIMARY OUTCOMES:
Number of sites with Bleeding on Probing | Bleeding on Probing (BOP) will be recorded by a calibrated and blinded examiner at the baseline visit and at one, two, three, and six months after treatment.
  Evaluate the additional effect on bleeding on probing of one month application of 0.12% CHX or 0.05% CHX + 0.05% CPC following a professional mechanical plaque removal (PMPR) session for a clinical evaluation period of 6 months in patients undergoing supportive periodontal therapy (gingivitis with reduced periodontium).

SECONDARY OUTCOMES:
Oral microbiota changes | The subgingival samples will be collected at the baseline visit, at 1, 2, and 3 months
  The DNA from subgingival samples will be used to sequence the V3-V4 region of the 16S rRNA gene and will be analyzed using PCR (Polymerase Chain Reaction). The amplicons will be purified and sequenced.
Blood Pressure | The systemic systolic and diastolic blood pressure will be measured at baseline, 1 month, 2 months, 3 months and 6 months.
  The systemic systolic and diastolic blood pressure (mmHg) will be measured in duplicate at each follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Discepoli, DDS MSc PhD, Principal Investigator — Department of Medical Biotechnologies, University of Siena
Locations (1):
- AOUS, Siena, Italy